CLINICAL TRIAL: NCT05809986
Title: Ofatumumab in Portuguese Multiple Sclerosis Patients - an Observational Study
Status: Recruiting | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157GPT04
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: Relapsing Multiple Sclerosis; RMS; Ofatumumab; NIS; Portugal
MeSH Terms: interventions — ofatumumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Cohort 1: Early treatment arm: All patients who initiated Ofatumumab within 3 years after MS diagnosis (can be treatment-naive or switch).
  Interventions: Other: Ofatumumab
- Cohort 2: Late treatment arm: All patients who initiated Ofatumumab with more than 3 years of MS diagnosis.
  Interventions: Other: Ofatumumab

INTERVENTIONS:
Other: Ofatumumab — There is no treatment allocation. Ofatumumab will be prescribed by the physician as per locally approved label. No drug will be dispensed from Novartis
  Other Names: Kesimpta

SUMMARY:
This non-interventional study will compare the effect of Ofatumumab treatment between patients that began Ofatumumab within the 3 years after Multiple Sclerosis diagnosis and patients that began Ofatumumab with more than 3 years of Multiple Sclerosis diagnosis in a real-world setting in Portugal.

DETAILED DESCRIPTION:
This is a 2 cohort, multi-center, observational study carried out in Portugal that aims to describe the effectiveness of Ofatumumab in a setting of routine medical care. Primary data will be collected from Multiple Sclerosis patients who initiate Ofatumumab early and later in their disease (cohorts 1 and 2, respectively).

Data will be collected during 3 visits distributed over a maximum period of 24 months. Exceptionally, if the patient shows Expanded Disability Status Scale (EDSS) worsening in visit 2 or 3 (12 and 24 months after Ofatumumab initiation, respectively), there will be an additional visit 6±1 months after visit 2 or 3 for EDSS confirmation.

The study includes patients that have initiated Ofatumumab up to 12 months prior inclusion in the study OR Patients that are initiating Ofatumumab at the moment of study inclusion.

Patients in both cohorts will have to be treated with Ofatumumab for at least two years to compare No Evidence of Disease Activity (NEDA)-3 at 12 to 24 months, respectively.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, all the following inclusion criteria must be met:

* Patients aged 18 years or older
* Written informed consent obtained before participating in the study.
* Patient is willing and able to complete the assessments, including PRO questionnaires, as outlined in this study.
* Diagnosis of RMS per McDonald Criteria (2017) occurred prior to initiation of Ofatumumab.
* Treatment with Ofatumumab is in accordance with the Portuguese indication of Kesimpta® (i.e., treatment of adult patients with relapsing multiple sclerosis (RMS) with active disease defined by clinical or imaging features).
* Patients that have initiated Ofatumumab up to 12 M prior inclusion in the study OR Patients that are initiating Ofatumumab at the moment of study inclusion.

Exclusion Criteria:

To participate in the study, none of the following exclusion criteria must be met:

* Use of investigational drugs during the study, OR between Ofatumumab initiation and inclusion into the study, OR within 5 half-lives of investigational drug before Ofatumumab initiation, OR until the expected pharmacodynamic effect has returned to baseline, whichever is longer.
* Use of high efficacy therapy (including Ocrelizumab, Natalizumab, Mitoxantrone, Rituximab and Alemtuzumab) in both cohorts prior to the initiation of Ofatumumab.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include male and female patients (aged ≥ 18 years) with a documented diagnosis of RMS and with Ofatumumab treatment in line with the Portuguese label i.e., adult patients with active, relapsing forms of MS.
Sampling Method: Non-Probability Sample
Enrollment: 174 (Estimated)
Dates: Start 2023-11-27 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-15 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients demonstrating NEDA-3 | from month 12 up to month 24
  Proportion of patients demonstrating No Evidence of Disease Activity (NEDA)-3 (12-24 months) in both cohorts, respectively. NEDA-3 is defined by no confirmed Multiple Sclerosis relapse, no new or enlarging T2 lesions, no Gadolinium-positive T1 lesions, and no six-month confirmed disability worsening.

SECONDARY OUTCOMES:
Proportion of patients demonstrating no evidence of disease activity in individual components of NEDA-3 | 12-24 months
  Proportion of patients demonstrating no evidence of disease activity in individual components of NEDA-3 (12-24 months) in the overall population and in both cohorts.
Multiple Sclerosis Impact Scale Questionnaire (MSIS-29) | Baseline, Month 12, Month 24
  Treatment effect of Ofatumumab on the impact of multiple sclerosis as measured by MSIS-29 (baseline, 12 and 24 months) in the overall population and in both cohorts.
  MSIS-29 is a 29-item self-report measure with 20 items associated with a physical scale and 9 items with a psychological scale. Items ask about the impact of MS on day-to-day life in the past two weeks. All items have 4 response options. Each score domain is obtained by summing all individual items and transformed it to a -100 scale where high scores indicate worse health.
Fatigue Symptoms and Impacts Questionnaire - Relapsing Multiple Sclerosis (FSIQ-RMS) | Baseline, Month 12, Month 24
  Treatment effect of Ofatumumab on the impact of multiple sclerosis as measured by FSIQ-RMS (baseline, 12 and 24 months) in the overall population and in both cohorts.
  The FSIQ-RMS is a patient-reported outcome (PRO) instrument used to assess fatigue in patients with relapsing types of multiple sclerosis (RMS).It is a 20-item self-report measure with 7 items for MS-related symptoms of fatigue and 13 for fatigue-related impacts on several aspects of patients' lives. The impact of fatigue divides into 3 subdomains: physical, cognitive and emotional, and coping. The scores for fatigue and the subdomains of impact are standardized to a 0-100 scale using a scoring algorithm, with higher scores indicating more severe symptoms and impacts.
Treatment Satisfaction Questionnaire for Multiple Sclerosis (TSQM-9) | Month 12, Month 24
  Treatment satisfaction with Ofatumumab as measured by TSQM-9 (baseline, 12 and 24 months) in the overall population and in both cohorts.
  The TSQM-9 is a validated tool, widely used, to measure treatment satisfaction that will be applied in the context of this study regarding Ofatumumab. The TSQM-9 uses nine of the 14 TSQM Version 1.4 items, not including five questions related to side effects of medication, and comprises three scales: the effectiveness scale, the convenience scale and the global scale. The TSQM-9 domain scores range from 0 to 100 with higher scores representing higher satisfaction on that domain.
Proportion of patients permanently discontinuing Ofatumumab during the study | up to month 24
  Proportion of patients permanently discontinuing Ofatumumab during the study, and reasons for discontinuation in the overall population and in both cohorts
Proportion of patients demonstrating NEDA-3 in the overall population. | 12-24 months
  Proportion of patients demonstrating NEDA-3 in the overall population.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (8):
- Portugal (8):
  - Novartis Investigative Site, Amadora
  - Novartis Investigative Site, Guimarães
  - Novartis Investigative Site, Leiria
  - Novartis Investigative Site, Lisbon
  - Novartis Investigative Site, Matosinhos Municipality
  - Novartis Investigative Site, Ponte de Lima
  - Novartis Investigative Site, Porto
  - Novartis Investigative Site, Setúbal

IPD SHARING:
Plan to Share IPD: No